CLINICAL TRIAL: NCT03020719
Title: A Multi Center Placebo Controlled Double Blind Randomized Study Evaluating the Role of Oral Glutathione on Growth Parameters in Children With Cystic Fibrosis
Brief Title: The Role of Oral Glutathione on Growth Parameters in Children With Cystic Fibrosis
Acronym: GROW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GROW-IP-16
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Cystic Fibrosis
Keywords: Growth Parameters; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Glutathione

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Glutathione (Experimental): Oral Glutathione oral powder at 65mg/kg/day
  Interventions: Drug: Oral Glutathione
- Placebo (Placebo Comparator): Placebo oral powder at 65mg/kg/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Glutathione — Oral Glutathione oral powder
  Other Names: GSH
  Arms: Oral Glutathione
Drug: Placebo — Placebo oral powder
  Other Names: Inactive powder
  Arms: Placebo

SUMMARY:
The purpose of this randomized, placebo-controlled (Phase II) study will be to further evaluate the effects of oral glutathione on growth in children with CF.

DETAILED DESCRIPTION:
a prospective, multi-center, randomized, placebocontrolled, double-blind, Phase II clinical trial. Approximately sixty pancreatic insufficient (PI) subjects with CF who are ≥ 2 and < 11 years of age, will be enrolled to receive either L-Glutathione Reduced (GSH) or placebo given orally (tid) for 24 weeks. Each subject will be seen for four study visits: Visit 1 (Screening), Visit 2 (Baseline/Randomization, Day 0), Visit 3 (Week 12) and Visit 4 (Week 24). At Visit 2, subjects will be randomized to receive either active treatment or placebo. Visit 1 and 2 may be combined if subject meets eligibility requirements and a fecal specimen is collected prior to dosing. Safety and clinical outcomes will be assessed throughout the study. Assessment of inflammatory and other bio-markers in blood and fecal specimens will be performed at Visits 2 and 4

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 2 and < 11 years of age at Visit 1
2. Documentation of a CF diagnosis as evidenced by the following criteria: Sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test (QPIT) AND Two well-characterized mutations in the cystic fibrosis transmembrane conductive regulator (CFTR) gene
3. Weight-for-age between the 10th and 50th percentiles at Screening (Visit 1) (using the Center for Disease Control (CDC) reference equations)
4. Current chronic use, greater than 8 weeks before Day 0, of pancreatic enzyme replacement therapy (PERT) for management of pancreatic insufficiency
5. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability to comply with the requirements of the study
6. Clinically stable with no significant changes in health status within 2 weeks prior to Day 0

Exclusion Criteria:

* 1. Intestinal obstruction or gastrointestinal surgery within the 6 months prior to Day 0 2. History of diabetes, Crohn's disease, celiac disease, or bowel resection 3. Use of either oral or inhaled GSH or N-acetyl cysteine within the 4 months prior to Screening (Visit 1) 4. Known hypersensitivity to oral glutathione or lactose 5. Initiation of any new chronic therapy (e.g., ibuprofen, hypertonic saline, azithromycin, Pulmozyme, Cayston TOBI Kalydeco,Orkambi, Proton Pump Inhibitor, Histamine H-2 Blocker [PPI/H2-blocker], Miralax® , PERT, dietary supplementation, probiotics) within the 4 weeks prior to Day 0 6. Changes in the amount of proprietary dietary supplement formulas (e.g., Scandishakes, Boost, Pediasure, or homemade formula) given (oral or gastrostomy tube) within the 4 weeks prior to Day 0 7. Use of antibiotics (oral, IV, or inhaled) for acute symptoms within the 2 weeks prior to Day 0 8. Use of oral steroids within the 4 weeks prior to Day 0 9. Active treatment for nontuberculous mycobacteria (NTM) at Day 0 10. Active treatment for allergic bronchopulmonary aspergillosis (ABPA) at Day 0 11. Administration of any investigational drug within the 30 days prior to Day 0 12. Sibling who received study drug as part of this study 13. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Schwarzenberg, MD, Principal Investigator — University of Minnesota; Molly Bozic, MD, Principal Investigator — Indiana University School of Medicine Riley Hospital
Locations (18):
- United States (18):
  - Childrens Hospital Colorado, Aurora, Colorado
  - Connecticut Childrens Medical Center, Hartford, Connecticut
  - Nemours Childrens Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Pensacola, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Riley Children's Hospital, Indianapolis, Indiana
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Helen DeVos Women and Childrens Center, Grand Rapids, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Women and Childrens Hospital of Buffalo, Buffalo, New York
  - Childrens Hospital of New York/Columbia University Medical Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Vermont Inc., Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Childrens Hospital of Milwaukee, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bozic M, Goss CH, Tirouvanziam RM, Baines A, Kloster M, Antoine L, Borowitz D, Schwarzenberg SJ; GROW study group. Oral Glutathione and Growth in Cystic Fibrosis: A Multicenter, Randomized, Placebo-controlled, Double-blind Trial. J Pediatr Gastroenterol Nutr. 2020 Dec;71(6):771-777. doi: 10.1097/MPG.0000000000002948. PMID 32960827

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Glutathione | Placebo
Started (Treated defined as having taken at least one dose of study drug.) | 30 | 30
Completed (Completed last study visit (Week 24).) | 30 | 28
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Glutathione | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (2.43) | 6 (2.87) | 6.1 (2.64)
Age, Customized [Count of Participants; unit: Participants]
  Age Distribution: < 6 years | 16 | 15 | 31
  Age Distribution: ≥ 6 years | 14 | 15 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 29 | 27 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 29 | 30 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Cystic Fibrosis (CF) Genotype [Count of Participants; unit: Participants] — Other refers to participants with either two known, non-F508 del CF mutations, or one known, non-F508 del CF mutation and one unidentified allele which has not been classified as a CF mutation. Unidentified refers to participants with 2 alleles that have not been classified as CF mutations.
  Participants
    Delta F508 Homozygous | 18 | 14 | 32
    Delta F508 Heterozygous | 9 | 13 | 22
    Other | 3 | 3 | 6
    Unidentified | 0 | 0 | 0
    Not Available | 0 | 0 | 0
Weight (Z-score) [Mean (Standard Deviation); unit: z-score] — Z-scores are derived from the 2000 Centers for Disease Control and Prevention growth charts for U.S. children. The reference population in these growth charts is children surveyed by the National Center for Health Statistics from 1963-65 to 1988-94. The Z-score indicates the number of standard deviations away from the mean of the reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
  z-score | -0.57 (0.33) | -0.53 (0.35) | -0.55 (0.34)
Weight-for-age Z-score Distribution [Count of Participants; unit: Participants] — Z-scores are derived from the 2000 Centers for Disease Control and Prevention growth charts for U.S. children. The reference population in these growth charts is children surveyed by the National Center for Health Statistics from 1963-65 to 1988-94. The Z-score indicates the number of standard deviations away from the mean of the reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
  Participants
    < -0.52 (equiv. to < 30th percentile) | 13 | 13 | 26
    ≥ -0.52 (equiv. to ≥ 30th percentile) | 17 | 17 | 34
Fecal Elastase [Count of Participants; unit: Participants] — Either historical fecal elastase or collected as part of the study.
  Participants
    < 200 mg/g | 30 | 30 | 60
    ≥ 200 mg/g | 0 | 0 | 0
    Not Available | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight-for-age Z-score
Description: Difference between the oral glutathione and placebo groups in the 24-week change from baseline in weight-for-age Z-score. Weight-for-age Z-scores are derived from the 2000 Centers for Disease Control and Prevention growth charts for U.S. children. The reference population in these growth charts is children surveyed by the National Center for Health Statistics from 1963-65 to 1988-94. The Z-score indicates the number of standard deviations away from the mean of the reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline to 24 weeks
Population: Include participants with weight-for-age Z-score measurements at Baseline, Week 12 and Week 24
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Oral Glutathione | Placebo
Number analyzed (Participants) | 30 | 28
Z-score | -0.018 [-0.124 to 0.087] | 0.045 [-0.073 to 0.163]
Statistical Analysis 1: Comparison: Oral Glutathione vs Placebo; Test type: Superiority; p = 0.2521, Mixed Models Analysis; Model adjusted for randomization strata: sex, baseline age (< 6 years, ≥ 6 years), and baseline weight-for-age z-score category (< -0.52, ≥ -0.52); Mean Difference (Final Values) = -0.081, 95% CI 2-sided [-0.221 to 0.059] — Model incorporates Week 12 weight-for-age z-score, assumes unstructured covariance for within-subject measurements, and includes a subject-level random intercept

2. Secondary Outcome: Change in Height-for-age Z-score
Description: Difference between the oral glutathione and placebo groups in the 24-week change from baseline in height-for-age Z-score. Height-for-age Z-scores are derived from the 2000 Centers for Disease Control and Prevention growth charts for U.S. children. The reference population in these growth charts is children surveyed by the National Center for Health Statistics from 1963-65 to 1988-94. The Z-score indicates the number of standard deviations away from the mean of the reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Oral Glutathione | Placebo
Number analyzed (Participants) | 30 | 28
Z-score | -0.04 (0.21) | 0.03 (0.16)
Statistical Analysis 1: Comparison: Oral Glutathione vs Placebo; Test type: Superiority; p = 0.0890, Mixed Models Analysis; Model adjusted for randomization strata: sex, baseline age (<6 years, ≥6 years), and baseline weight-for-age z-score category (< -0.52, ≥-0.52); Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.18 to 0.01] — Model incorporates Week 12 measurements, assumes unstructured covariance for within-subject measurements, and includes a subject-level random intercept

3. Secondary Outcome: Change in BMI-for-age Z-score
Description: Difference between the oral glutathione and placebo groups in the 24-week change from baseline in BMI-for-age Z-score. BMI-for-age Z-scores are derived from the 2000 Centers for Disease Control and Prevention growth charts for U.S. children. The reference population in these growth charts is children surveyed by the National Center for Health Statistics from 1963-65 to 1988-94. The Z-score indicates the number of standard deviations away from the mean of the reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Oral Glutathione | Placebo
Number analyzed (Participants) | 30 | 28
Z-score | -0.01 (0.48) | 0.04 (0.44)
Statistical Analysis 1: Comparison: Oral Glutathione vs Placebo; Test type: Superiority; p = 0.5730, Mixed Models Analysis; Model adjusted from randomization strata: sex, baseline age (<6 years, ≥6 years), and baseline weight-for-age z-score category (< -0.52, ≥-0.52); Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.28 to 0.15] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change in Fecal Calprotectin
Description: Difference between the oral glutathione and placebo groups in the 24-week change from baseline in fecal calprotectin.
Time Frame: Baseline to 24 weeks
Population: Include participants with fecal calprotectin measurements at Baseline and Week 24.
Measure: Mean (Standard Deviation); unit: log base 10 transformation of ug/g
Arm/Group | Oral Glutathione | Placebo
Number analyzed (Participants) | 29 | 26
log base 10 transformation of ug/g | 0.05 (0.55) | -0.05 (0.53)
Statistical Analysis 1: Comparison: Oral Glutathione vs Placebo; Test type: Superiority; p = 0.4259, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.17 to 0.40] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change in High-sensitivity C-reactive Protein (Hs-CRP)
Description: Difference between the oral glutathione and placebo groups in the 24-week change from baseline in hs-CRP.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Oral Glutathione | Placebo
Number analyzed (Participants) | 29 | 25
mg/L | -0.45 (3.4) | -0.04 (1.6)
Statistical Analysis 1: Comparison: Oral Glutathione vs Placebo; Test type: Superiority; p = 0.4666, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-2.06 to 0.96]

6. Secondary Outcome: Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: The number and percentage of participants with at least one event over the 24 week follow-up period.
Time Frame: Baseline to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Glutathione | Placebo
Number analyzed (Participants) | 30 | 30
Participants
  Adverse Events | 29 | 29
  Serious Adverse Events | 1 | 5
Statistical Analysis 1: Comparison: Oral Glutathione vs Placebo; Test type: Superiority; p = 1.0000, Fisher Exact; Difference in % of Participants with AE = 0.0, 95% CI 2-sided [-13.6 to 13.6] — 95% CI calculated using the Newcombe-Wilson method without continuity correction
Statistical Analysis 2: Comparison: Oral Glutathione vs Placebo; Test type: Superiority; p = 0.1945, Fisher Exact; Difference in % of Participants with SAE = -13.3, 95% CI 2-sided [-30.5 to 2.9] — 95% CI calculated using the Newcombe-Wilson method without continuity correction

7. Secondary Outcome: Rate of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Rate is defined as the number of events per participant follow-up month.
Time Frame: Baseline to 24 weeks
Measure: Number; unit: number of events/total follow-up months
Arm/Group | Oral Glutathione | Placebo
Number analyzed (Participants) | 30 | 30
number of events/total follow-up months
  Adverse Events | 0.89 | 0.74
  Serious Adverse Events | 0.01 | 0.05
Statistical Analysis 1: Comparison: Oral Glutathione vs Placebo; Rate Ratio for Adverse Events calculated using Poisson Regression with an offset for the log of follow-up time in months. The total number of follow-up months of all participants (not per participant) in the trial was as follows: in the GSH group was 179.22 and in the Placebo group was 177.19; Test type: Superiority; p = 0.1087, Poisson Regression; Rate Ratio = 1.21, 95% CI 2-sided [0.96 to 1.52]
Statistical Analysis 2: Comparison: Oral Glutathione vs Placebo; Rate Ratio for Serious Adverse Events calculated using Poisson Regression with an offset for the log of follow-up time in months. The total number of follow-up months of all participants (not per participant) in the trial was as follows: in the GSH group was 179.22 and in the Placebo group was 177.19; Test type: Superiority; p = 0.0122, Poisson Regression; Rate Ratio = 0.12, 95% CI 2-sided [0.01 to 0.67]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Oral Glutathione | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 5/30
Other Adverse Events (participants affected / at risk) | 29/30 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Glutathione (N=30) | Placebo (N=30)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infective pulmonary exacerbation of cystic fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Glutathione (N=30) | Placebo (N=30)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Steatorrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (9) | 6 (6)
Pyrexia (General disorders) | 8 (12) | 5 (6)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 6 (6) | 1 (1)
Sinusitis (Infections and infestations) | 6 (7) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 6 (8)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Pulmonary function test decreased (Investigations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 5 (5) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Clubbing (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (24) | 12 (14)
Infective pulmonary exacerbation of cystic fibrosis (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 9 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT03020719/SAP_000.pdf
  • Study Protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT03020719/Prot_001.pdf